CLINICAL TRIAL: NCT02108964
Title: A Phase I/II, Multicenter, Open-label Study of EGFRmut-TKI EGF816, Administered Orally in Adult Patients With EGFRmut Solid Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEGF816X2101; 2013-004482-14 (EudraCT Number)
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Advanced Non-small Cell Lung Cancer
Keywords: NSCLC; Non-small Cell Lung Cancer EGFRmut; EGFR TKIs (EGF816); acquired T790M mutation; de novo T790M mutation; EGFR TKI activating mutation (i.e. L858R or ex19del); Treatment naive advanced NSCLC with EGFR activating mutations; Locally advanced NSCLC (Stage IIIB NSCLC not amenable to definitive multi-modality therapy including surgery); Metastatic NSCLC refers to Stage IV NSCLC; 1st line
MeSH Terms: interventions — nazartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I part (Experimental): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations will be administered escalated doses of EGF816 orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study. The starting dose for the Phase I part first cohort of patients will be 75 mg once per day capsule.
  Interventions: Drug: EGF816
- Phase II part (Experimental): Treatment naïve participants with locally advanced or metastatic NSCLC harboring EGFR mutations will be administered with EGF816 at RP2D during Phase II part of the study.
  Interventions: Drug: EGF816

INTERVENTIONS:
Drug: EGF816 — EGF816 will be dosed once daily. On the first day of each treatment cycle, the patient receives an adequate drug supply for self-administration at home. The investigator will instruct the patient to take EGF816 exactly as prescribed.
  Other Names: Nazartinib

SUMMARY:
This is a Phase I/II, multi-center, open-label study, composed with a Phase I part (dose-escalation phase) followed by a Phase II part (expansion phase).

The dose escalation phase was designed to determine as primary objective the maximum tolerated dose (MTD) or recommended Phase II dose (RP2D) of EGF816 monotherapy in adult subjects with locally advanced (stage IIIB) or metastatic (stage IV) NSCLC harboring specific EGFR mutations. Patients may have or not have received prior lines of antineoplastic therapy. An adaptive Bayesian Logistic Regression Model (BLRM) employing the escalation with overdose control (EWOC) principle will be used during the dose escalation part for dose level selection and MTD recommendation. The primary objective of the Phase II part is to estimate antitumor activity of EGF816 as measured by overall response rate (ORR) determined by Blinded Independent Review Committee (BIRC) assessment in accordance to RECIST 1.1.

DETAILED DESCRIPTION:
Following completion of screening procedures and confirmation of patient eligibility, the participants are enrolled in the study. The study treatment begin on Cycle 1, Day 1 with the first administration of EGF816. A treatment cycle is defined as 28 days. Oral EGF816 is administered once daily on a continuous schedule until patient experiences unacceptable toxicity, progressive disease (PD), and/or treatment is discontinued at the discretion of the investigator, patient withdrawal of consent, or due to any other reasons. Treatment with EGF816 may be continued beyond RECIST 1.1 defined PD, if, in the judgment of the investigator, there is evidence of clinical benefit and the patient wishes to continue with the study treatment.

ELIGIBILITY:
Inclusion Criteria: (For all patients unless otherwise specified)

* Histologically or cytologically confirmed locally advanced (stage IIIB not amenable to definitive multi-modality therapy including surgery) or metastatic (stage IV) EGFR mutant NSCLC.
* Patients with controlled brain metastases
* ECOG performance status: Phase I part: 0, 1, or 2; Phase II part: 0 or 1
* Presence of at least one measurable lesion according to RECIST 1.1 per investigator assessment
* Patients who are either Hepatitis B surface antigen (HBsAg) positive or hepatitis B virus (HBV)-DNA positive must be willing and able to take antiviral therapy 1-2 weeks prior to 1st dose of EGF816 treatment and continue on antiviral therapy for at least 4 weeks after the last dose of EGF816
* Patients must have negative hepatitis C antibody (HCV-Ab) or positive HCV-Ab but undetectable level of HCV-RNA. Note: patients with detectable HCV-RNA are not eligible for the study.
* For Phase I: patients must have failed no more than 3 lines of any systemic antineoplastic therapy for advanced NSCLC, including EGFR-TKI
* For Phase II: patients must be naïve from any systemic antineoplastic therapy in the advanced setting. Patients who have failed no more than 1 cycle of systemic antineoplastic therapy in the advanced setting are allowed.

Exclusion criteria: (For all patients unless otherwise specified)

* Patients with a history or presence of interstitial lung disease (ILD) or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e. affecting activities of daily living or requiring therapeutic intervention)
* Presence or history of another malignancy
* Undergone a bone marrow or solid organ transplant
* Known history of human immunodeficiency virus (HIV) seropositivity
* Patients receiving concomitant immunosuppressive agents or chronic corticosteroids use at the time of study entry except for control of brain metastases, topical applications, inhaled sprays, eye drops or local injections
* Patients with clinically significant, uncontrolled heart disease
* Any prior therapies ≤ 4 weeks prior to the first dose of study treatment
* Patients who are receiving treatment with medications that are known to be strong inhibitors or inducers of CYP3A4/5 and cannot be discontinued 1 week prior to the start of EGF816 treatment and for the duration of the study.
* Patients who have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of EGF816
* Patients who are receiving treatment with any enzyme-inducing anticonvulsant that cannot be discontinued at least 1 week before first dose of study treatment, and for the duration of the study
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception
* Sexually active males unless they use a condom during intercourse while taking drug and for 3 months after stopping treatment

Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (2):
  - Massachusetts General Hospital Mass General, Boston, Massachusetts
  - Memorial Sloan Kettering Oncology Department, New York, New York
- Novartis Investigative Site, Toronto, Ontario, Canada
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
- Japan (2):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
- Novartis Investigative Site, Zoetermeer, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Tan DSW, Kim SW, Ponce Aix S, Sequist LV, Smit EF, Yang JCH, Hida T, Toyozawa R, Felip E, Wolf J, Grohe C, Leighl NB, Riely G, Cui X, Zou M, Ghebremariam S, O'Sullivan-Djentuh L, Belli R, Giovannini M, Kim DW. Nazartinib for treatment-naive EGFR-mutant non-small cell lung cancer: Results of a phase 2, single-arm, open-label study. Eur J Cancer. 2022 Sep;172:276-286. doi: 10.1016/j.ejca.2022.05.023. Epub 2022 Jul 7. PMID 35810553
- [Derived] Tan DS, Leighl NB, Riely GJ, Yang JC, Sequist LV, Wolf J, Seto T, Felip E, Aix SP, Jonnaert M, Pan C, Tan EY, Ko J, Moody SE, Kim DW. Safety and efficacy of nazartinib (EGF816) in adults with EGFR-mutant non-small-cell lung carcinoma: a multicentre, open-label, phase 1 study. Lancet Respir Med. 2020 Jun;8(6):561-572. doi: 10.1016/S2213-2600(19)30267-X. Epub 2020 Jan 15. PMID 31954624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a 2-part study conducted in 14 investigative sites in 9 countries: Phase I part (dose-escalation) and Phase II part (dose expansion)
Pre-assignment Details: 370 subjects were screened for eligibility during the 28 days prior to starting study treatment on Cycle 1 Day 1 (C1D1). The eligibility assessments were performed and ensured that all inclusion and exclusion criteria were satisfied
Groups:
- EGF816 75 mg (Phase I Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 75 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF816 100 mg (Phase I Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 100 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF816 150 mg (Phase I Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 150 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF816 200 mg (Phase I Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 200 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF816 225 mg (Phase I Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 225 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF816 300 mg (Phase I Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 300 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF816 350 mg (Phase I Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 350 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF816 150 mg (Phase II Part): Treatment naïve participants with locally advanced or metastatic NSCLC harboring EGFR mutations were administered with 150 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase II part of the study.
Period: Overall Study
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part) | EGF816 150 mg (Phase II Part)
Started | 17 | 38 | 73 | 8 | 28 | 5 | 11 | 45
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 17 | 38 | 73 | 8 | 28 | 5 | 11 | 45
Not completed — Progressive disease | 15 | 31 | 54 | 7 | 20 | 4 | 6 | 33
Not completed — Physician Decision | 1 | 5 | 7 | 1 | 2 | 1 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 4 | 0 | 1 | 0 | 3 | 2
Not completed — Death | 1 | 1 | 4 | 0 | 3 | 0 | 0 | 2
Not completed — Subject/Guardian decision | 0 | 1 | 4 | 0 | 2 | 0 | 1 | 2
Not completed — Study terminated by Sponsor: remaining participants benefiting from drug were transitioned to PSDS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The full analysis set (FAS) includes all subjects who received at least one dose of EGF816.
Groups:
- Total: Total of all reporting groups
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part) | EGF816 150 mg (Phase II Part) | Total
Number analyzed (Participants) | 17 | 38 | 73 | 8 | 28 | 5 | 11 | 45 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 23 | 47 | 6 | 15 | 2 | 7 | 23 | 133
  >=65 years | 7 | 15 | 26 | 2 | 13 | 3 | 4 | 22 | 92
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 23 | 50 | 7 | 13 | 3 | 7 | 27 | 143
  Male | 4 | 15 | 23 | 1 | 15 | 2 | 4 | 18 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13 | 22 | 44 | 6 | 21 | 4 | 9 | 28 | 147
  Caucasian | 2 | 14 | 24 | 2 | 7 | 1 | 2 | 17 | 69
  Unknown | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 7
  Black | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) (Phase I Part)
Description: Number of participants with DLTs during the first 28 days of therapy. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle of treatment with EGF816 and meets any of the criteria described in the protocol. A participant with multiple occurrences of DLTs under one treatment is counted only once.
Time Frame: First 28 days of dosing
Population: Dose-determining set (DDS) including all patients who received at least one dose of EGF816 in the dose escalation phase who had met the minimum safety evaluation requirements (observed for ≥ 28 days following the first dose) and the minimum exposure criterion (at least 75% of the planned doses of EGF816) or discontinue earlier due to DLTs
Measure: Count of Participants; unit: Participants
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part)
Number analyzed (Participants) | 16 | 38 | 69 | 7 | 23 | 2 | 9
Participants | 0 | 0 | 2 | 0 | 1 | 0 | 3

2. Primary Outcome: Overall Response Rate (ORR) by Blinded Independent Review Committee (BIRC) (Phase II Part)
Description: ORR is defined as the percentage of patients with a best overall response of complete response (CR) or partial response (PR) determined by BIRC assessment in accordance to Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
Time Frame: From baseline up to 64 weeks
Population: Full Analysis Set (FAS) including participants who received at least one dose of EGF816
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 45
Percentage of participants | 64.4 [48.80 to 78.10]

3. Secondary Outcome: Progression-free Survival (PFS) by Investigator Assessment (Phase I & Phase II Parts)
Description: PFS is defined as time from date of first dose of study treatment to date of first documented disease progression or death due to any cause determined by Investigator assessment in accordance to RECIST 1.1
Time Frame: At least 24 weeks up to approx. 9 years
Population: Full Analysis Set (FAS) including participants who received at least one dose of EGF816
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part) | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 12 | 34 | 68 | 8 | 24 | 5 | 11 | 45
Months | 6.3 [1.54 to 47.80] | 12.1 [7.16 to 16.56] | 7.4 [5.32 to 9.59] | 13.7 [3.52 to 27.47] | 11.1 [7.23 to 23.49] | 11.8 [5.62 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | 11.0 [0.43 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | 18.2 [11.04 to 30.16]

4. Secondary Outcome: Duration of Response (DOR) by Investigator Assessment (Phase I & II Parts)
Description: DOR is defined as the time from first documented response (PR or CR) to the date of first documented disease progression or death due to any cause determined by Investigator assessment in accordance to RECIST 1.1
Time Frame: At least 24 weeks up to approx. 9 years
Population: Full Analysis Set (FAS) including participants who received at least one dose of EGF816
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part) | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 5 | 17 | 34 | 5 | 15 | 3 | 4 | 29
Months | 46.2 [3.68 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | 11.3 [7.39 to 23.79] | 7.9 [7.39 to 11.04] | 14.9 [9.20 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | 16.5 [5.52 to 29.63] | 10.2 [9.33 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | 17.5 [7.56 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | 20.3 [11.01 to 34.89]

5. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) of EGF816 and Metabolite LMI258 (Phase I & Phase II Part)
Description: To characterize the PK properties of EGF816 and metabolite LMI258, Cmax will be calculated (Phase I & II parts).
  Cmax is maximum (peak) observed plasma drug concentration (mass x volume-1).
Time Frame: Cycle (C) 1 Day (D) 1 (pre-dose and 0.5,1,2,3,4,6,8,12 and 24 hours (hrs) post-dose), C1D15 (pre-dose and 0.5,1,2,3,4,6,8,12 and 24 hrs post-dose) (for Phase I part only) and C2D1 (pre-dose and 0.5,1,2,3,4,6,8,12 and 24 hrs post-dose).
Population: Pharmacokinetics Analysis Set (PAS) The PAS consists of all subjects who received at least one dose of EGF816 and have at least one evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part) | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 17 | 38 | 72 | 8 | 28 | 5 | 11 | 45
ng/mL
  EFG816: Cycle (C) 1 Day (D) 1: number analyzed (Participants) | 17 | 36 | 69 | 8 | 28 | 5 | 11 | 45
  EFG816: Cycle (C) 1 Day (D) 1 | 333 (64.9) | 301 (81.8) | 541 (53.2) | 641 (60.2) | 935 (66.1) | 1070 (58.3) | 1190 (50.0) | 471 (41.2)
  EFG816: C1D15: number analyzed (Participants) | 14 | 36 | 63 | 7 | 21 | 1 | 6 | 0
  EFG816: C1D15 | 402 (62.3) | 477 (53.0) | 765 (50.1) | 939 (45.4) | 1320 (46.0) | 2670 (NA) — NA = Geo CV% could not be reached due to the low number of participants analyzed. | 1530 (23.5) |
  EFG816: C2D1: number analyzed (Participants) | 12 | 24 | 59 | 7 | 20 | 3 | 9 | 26
  EFG816: C2D1 | 348 (43.4) | 426 (50.1) | 767 (46.7) | 938 (53.9) | 1270 (61.0) | 1700 (41.3) | 1270 (30.4) | 648 (50.9)
  LMI258: C1D1: number analyzed (Participants) | 17 | 36 | 68 | 8 | 28 | 5 | 11 | 38
  LMI258: C1D1 | 14.1 (174.8) | 11.4 (76.1) | 25.2 (61.7) | 30.9 (64.6) | 42.0 (63.1) | 62.2 (40.5) | 52.7 (42.1) | 24.3 (46.6)
  LMI258: C1D15: number analyzed (Participants) | 13 | 34 | 61 | 7 | 20 | 1 | 5 | 0
  LMI258: C1D15 | 31.2 (94.7) | 34.1 (81.8) | 72.2 (64.0) | 113 (54.1) | 131 (56.8) | 292 (NA) — NA = NA = Geo CV% could not be reached due to the low number of participants analyzed. | 164 (22.7) |
  LMI258: C2D1: number analyzed (Participants) | 10 | 30 | 54 | 6 | 16 | 3 | 7 | 13
  LMI258: C2D1 | 23.9 (59.5) | 32.4 (76.0) | 81.4 (55.4) | 114 (75.1) | 101 (72.8) | 142 (55.1) | 116 (68.7) | 62.5 (60.7)

6. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of EGF816 and Metabolite LMI258 (Phase I & Phase II Part). Tmax is the Time to Reach Maximum (Peak) Plasma Drug Concentration (Time).
Description: To characterize the PK properties of EGF816 and metabolite LMI258, Tmax will be calculated (Phase I & II parts). Tmax is the time to reach maximum (peak) plasma drug concentration (time).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (hr)
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part) | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 17 | 38 | 69 | 8 | 28 | 5 | 11 | 43
hour (hr)
  EFG816: Cycle (C) 1 Day (D) 1: number analyzed (Participants) | 17 | 36 | 69 | 8 | 28 | 5 | 11 | 43
  EFG816: Cycle (C) 1 Day (D) 1 | 2.83 (63.0) | 3.24 (42.7) | 2.74 (54.7) | 3.66 (74.1) | 2.64 (64.9) | 3.37 (41.0) | 3.45 (22.4) | 2.81 (43.4)
  EFG816: C1D15: number analyzed (Participants) | 14 | 36 | 63 | 7 | 21 | 1 | 6 | 0
  EFG816: C1D15 | 2.91 (57.7) | 2.75 (75.8) | 3.11 (46.4) | 3.52 (44.3) | 3.46 (36.1) | 6.08 (NA) — NA = Geo CV% could not be reached due to the low number of participants analyzed. | 4.45 (35.4) |
  EFG816: C2D1: number analyzed (Participants) | 12 | 34 | 59 | 7 | 20 | 3 | 9 | 26
  EFG816: C2D1 | 3.13 (44.7) | 2.81 (49.0) | 3.14 (54.0) | 3.53 (35.3) | 3.17 (38.2) | 2.99 (0.6) | 3.97 (44.1) | 3.48 (52.7)
  LMI258: C1D1: number analyzed (Participants) | 17 | 36 | 68 | 8 | 28 | 5 | 11 | 38
  LMI258: C1D1 | 2.54 (65.7) | 3.14 (43.6) | 2.78 (65.2) | 3.19 (73.6) | 2.99 (71.4) | 3.37 (41.5) | 3.53 (31.8) | 2.70 (43.3)
  LMI258: C1D15: number analyzed (Participants) | 13 | 34 | 61 | 7 | 20 | 1 | 5 | 0
  LMI258: C1D15 | 2.89 (55.1) | 2.76 (63.8) | 3.32 (54.7) | 4.05 (32.6) | 4.03 (38.7) | 7.12 (NA) — NA = Geo CV% could not be reached due to the low number of participants analyzed. | 4.54 (39.3) |
  LMI258: C2D1: number analyzed (Participants) | 10 | 33 | 57 | 7 | 19 | 3 | 8 | 13
  LMI258: C2D1 | 3.38 (64.7) | 3.04 (57.6) | 3.43 (55.0) | 5.00 (56.1) | 3.26 (46.6) | 3.77 (42.4) | 4.13 (47.8) | 3.92 (45.5)

7. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau (AUCtau) of EGF816 and Metabolite LMI258 (Phase I & Phase II Part)
Description: To characterize the PK properties of EGF816 and metabolite LMI258, AUCtau will be calculated (Phase I & II parts). AUCtau is the AUC calculated to the end of a dosing interval (tau) (amount x time x volume-1).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part) | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 17 | 38 | 72 | 8 | 28 | 5 | 11 | 45
ng*hr/mL
  EFG816: Cycle (C) 1 Day (D) 1: number analyzed (Participants) | 16 | 35 | 66 | 8 | 26 | 5 | 11 | 41
  EFG816: Cycle (C) 1 Day (D) 1 | 4340 (68.2) | 4000 (83.1) | 6880 (53.3) | 8310 (51.2) | 12100 (64.7) | 15000 (61.0) | 16900 (51.0) | 5720 (42.7)
  EFG816: C1D15: number analyzed (Participants) | 13 | 31 | 57 | 7 | 18 | 1 | 5 | 0
  EFG816: C1D15 | 6370 (61.1) | 6770 (66.0) | 11300 (53.2) | 13500 (44.1) | 20300 (54.6) | 51200 (NA) — NA = Geo CV% could not be reached due to the low number of participants analyzed. | 25700 (26.1) |
  EFG816: C2D1: number analyzed (Participants) | 12 | 30 | 56 | 6 | 17 | 3 | 7 | 25
  EFG816: C2D1 | 5670 (44.7) | 6150 (58.6) | 11800 (50.3) | 15800 (10.6) | 18600 (66.5) | 26100 (53.0) | 22300 (19.0) | 9830 (51.3)
  LMI258: C1D1: number analyzed (Participants) | 15 | 33 | 65 | 8 | 26 | 5 | 11 | 37
  LMI258: C1D1 | 182 (56.8) | 162 (78.0) | 330 (62.1) | 424 (56.0) | 559 (62.4) | 859 (50.0) | 810 (47.0) | 291 (45.3)
  LMI258: C1D15: number analyzed (Participants) | 13 | 31 | 57 | 7 | 19 | 1 | 5 | 0
  LMI258: C1D15 | 466 (82.1) | 523 (111.1) | 1170 (69.5) | 1810 (58.6) | 2460 (65.2) | 5940 (NA) — NA = Geo CV% could not be reached due to the low number of participants analyzed. | 3420 (45.6) |
  LMI258: C2D1: number analyzed (Participants) | 10 | 30 | 54 | 6 | 16 | 3 | 7 | 13
  LMI258: C2D1 | 402 (65.7) | 499 (97.7) | 1380 (58.6) | 2340 (45.2) | 1760 (90.3) | 2360 (65.9) | 2820 (34.8) | 1060 (67.7)

8. Secondary Outcome: Percentage Change From Baseline in H-score for Immunohistochemistry (IHC) Biomarkers From Tumor Tissue Samples (Phase I Part)
Description: Changes in EGFR signaling pathway of newly obtained tumor samples following EGF816 treatment were evaluated by IHC of three pharmacodynamics (PD) biomarkers: p-EGFR, p-AKT and p-ERK. The assigned H-score semi-quantitatively assessed the expression level of these protein markers and their phosphorylated forms.
Time Frame: Baseline and Cycle 1 Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part) | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 2 | 5 | 10 | 4 | 9 | 2 | 4 | 0
percentage change
  Pharmacodynamics (PD) parameter: P_AKT: % Change from baseline in H-Score: number analyzed (Participants) | 1 | 5 | 10 | 4 | 9 | 2 | 4 | 0
  Pharmacodynamics (PD) parameter: P_AKT: % Change from baseline in H-Score | -10.0 (NA) — NA = SD could not be calculated due to the low number of participants analyzed. | -39.0 (78.2) | -31.8 (47.7) | 3.5 (14.5) | 16.1 (65.3) | -2.5 (3.5) | -51.3 (71.9) |
  PD parameter: p-EGFR: % Change from baseline in H-Score: number analyzed (Participants) | 1 | 5 | 10 | 4 | 9 | 2 | 4 | 0
  PD parameter: p-EGFR: % Change from baseline in H-Score | -165.0 (NA) — NA = SD could not be calculated due to the low number of participants analyzed. | -21.8 (43.9) | -19.5 (34.7) | -38.8 (50.1) | 2.2 (23.7) | -32.5 (38.9) | -12.5 (18.9) |
  PD parameter: p-ERK: % Change from baseline in H-Score: number analyzed (Participants) | 1 | 5 | 10 | 4 | 8 | 2 | 4 | 0
  PD parameter: p-ERK: % Change from baseline in H-Score | -60.0 (NA) — NA = SD could not be calculated due to the low number of participants analyzed. | -113.4 (84.2) | -2.4 (128.3) | 33.5 (86.7) | 8.8 (68.0) | -65.0 (35.4) | -1.3 (46.6) |

9. Secondary Outcome: Overall Response Rate (ORR) by Investigator Assessment (Phase I & II Parts)
Description: ORR is defined as percentage of patients with best overall response of partial response (PR)+ complete response (CR) determined by Investigator assessment in accordance to RECIST 1.1
Time Frame: At least 24 weeks up to approx. 4 years
Population: Full Analysis Set (FAS) including participants who received at least one dose of EGF816 and who had a response.
Measure: Number; unit: Percentage of participants
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part) | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 12 | 34 | 68 | 8 | 24 | 5 | 11 | 45
Percentage of participants | 41.7 | 50.0 | 50.0 | 62.5 | 62.5 | 60.0 | 36.4 | 55.6

10. Secondary Outcome: Disease Control Rate (DCR) by Investigator Assessment (Phase I & II Parts)
Description: DCR is defined as the proportion of patients with best overall response of CR, PR, or SD determined by Investigator assessment in accordance to RECIST 1.1
Time Frame: At least 24 weeks up to approx. 4 years
Population: Full Analysis Set (FAS) including participants who received at least one dose of EGF816 and who had a response.
Measure: Number; unit: Percentage of participants
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part) | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 12 | 34 | 68 | 8 | 24 | 5 | 11 | 45
Percentage of participants | 83.3 | 97.1 | 83.3 | 100.0 | 95.8 | 100.0 | 72.7 | 91.1

11. Secondary Outcome: Time to Response (TTR) by Investigator Assessment (Phase I & II Parts)
Description: TTR is defined as the time from the date of the first dose to the date of first documented response (CR or PR) determined by Investigator assessment in accordance to RECIST 1.1
Time Frame: At least 24 weeks up to approx. 9 years
Population: Full Analysis Set (FAS) including participants who received at least one dose of EGF816 and who had a response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part) | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 12 | 34 | 68 | 8 | 24 | 5 | 11 | 45
Months | NA [1.64 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | 5.5 [1.81 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | 11.6 [1.87 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | 4.5 [1.64 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | 1.9 [1.68 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | 1.7 [1.61 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | NA [1.64 to NA] — NA = the upper limit of CI was not reached as there were not enough events observed | 1.9 [1.84 to 7.16]

12. Secondary Outcome: Number of Participants With Dose Interruptions and Dose Reductions (Phase I & II Parts)
Description: Assessment of the tolerability of EGF816 will be performed continuously during the treatment phase
Time Frame: At least 24 weeks up to approx. 9 years
Population: Safety Set: The Safety Set includes all subjects who received at least one dose of EGF816.
Measure: Count of Participants; unit: Participants
Arm/Group | EGF816 75 mg (Phase I Part) | EGF816 100 mg (Phase I Part) | EGF816 150 mg (Phase I Part) | EGF816 200 mg (Phase I Part) | EGF816 225 mg (Phase I Part) | EGF816 300 mg (Phase I Part) | EGF816 350 mg (Phase I Part) | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 17 | 38 | 73 | 8 | 28 | 5 | 11 | 45
Participants
  Participants with any dose Interruption | 3 | 17 | 35 | 5 | 20 | 5 | 6 | 19
  Participants with at least one dose reductions | 0 | 1 | 9 | 1 | 17 | 4 | 6 | 9

13. Secondary Outcome: Duration of Response (DOR) by BIRC (Phase II Part)
Description: DOR is defined as the time from first documented response (PR or CR) to the date of first documented disease progression or death due to any cause determined by BIRC in accordance to RECIST 1.1
Time Frame: At least 24 weeks up to approx. 9 years
Population: Full Analysis Set (FAS) including participants who received at least one dose of EGF816 and who had a response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 30
Months | 18.6 [14.88 to 31.41]

14. Secondary Outcome: Disease Control Rate (DCR) by BIRC (Phase II Part)
Description: DCR is defined as the percentage of patients with best overall response of CR, PR, or SD determined by BIRC in accordance to RECIST 1.1
Time Frame: At least 24 weeks up to approx. 9 years
Population: Full Analysis Set (FAS) including participants who received at least one dose of EGF816
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 45
Percentage of participants | 93.3 [81.70 to 98.60]

15. Secondary Outcome: Progression-Free Survival (PFS) by BIRC (Phase II Part)
Description: PFS is defined as time from date of first dose of study treatment to date of first documented disease progression or death due to any cause determined by BIRC in accordance to RECIST 1.1
Time Frame: At least 24 weeks up to approx. 9 years
Population: Full Analysis Set (FAS) including participants who received at least one dose of EGF816
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 45
months | 18.9 [14.75 to 29.44]

16. Secondary Outcome: Time to Response (TTR) by BIRC (Phase II Part)
Description: TTR is defined as as the time from the date of first dose of study treatment to the date of first documented response (CR or PR) determined by by BIRC in accordance to RECIST 1.1
Time Frame: At least 24 weeks up to approx. 9 years
Population: Full Analysis Set (FAS) including participants who received at least one dose of EGF816
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 45
Months | 48.3 [22.93 to 58.84]

17. Secondary Outcome: Overall Survival (OS) (Phase II Part)
Description: OS is defined as the time from first dose of the study treatment to the date of death due to any cause.
Time Frame: At least 24 weeks up to approx. 9 years
Population: Full Analysis Set (FAS) including participants who received at least one dose of EGF816
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGF816 150 mg (Phase II Part)
Number analyzed (Participants) | 45
Months | 48.3 [22.93 to 58.84]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are collected from first dose of study treatment until end of study treatment plus 30 days post treatment. AEs reported in this record are from first dose of study treatment until 30 days after end of treatment, approx. 9 years.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Groups:
- EGF816 75 mg (Phase l Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 75 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF816 100 mg (Phase l Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 100 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF816 150 mg (Phase l Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 150 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF816 200 mg (Phase l Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 200 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF8166 225 mg (Phase l Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 225 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF816 300 mg (Phase l Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 300 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- EGF816 350 mg (Phase l Part): Participants with locally advanced or metastatic NSCLC harboring specific EGFR mutations were administered with EGF816 350 mg orally once a day as continuous daily dosing in each cycle (of 28 days) during Phase I part of the study.
- All Subjects: All subjects in the phase l and phase ll parts of the study.
Arm/Group | EGF816 75 mg (Phase l Part) | EGF816 100 mg (Phase l Part) | EGF816 150 mg (Phase l Part) | EGF816 200 mg (Phase l Part) | EGF8166 225 mg (Phase l Part) | EGF816 300 mg (Phase l Part) | EGF816 350 mg (Phase l Part) | EGF816 150 mg (Phase II Part) | All Subjects
All-Cause Mortality (participants affected / at risk) | 3/17 | 1/38 | 13/73 | 0/8 | 7/28 | 0/5 | 1/11 | 6/45 | 31/225
Serious Adverse Events (participants affected / at risk) | 7/17 | 11/38 | 40/73 | 2/8 | 16/28 | 4/5 | 5/11 | 22/45 | 107/225
Other Adverse Events (participants affected / at risk) | 17/17 | 36/38 | 73/73 | 8/8 | 28/28 | 5/5 | 11/11 | 42/45 | 220/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EGF816 75 mg (Phase l Part) (N=17) | EGF816 100 mg (Phase l Part) (N=38) | EGF816 150 mg (Phase l Part) (N=73) | EGF816 200 mg (Phase l Part) (N=8) | EGF8166 225 mg (Phase l Part) (N=28) | EGF816 300 mg (Phase l Part) (N=5) | EGF816 350 mg (Phase l Part) (N=11) | EGF816 150 mg (Phase II Part) (N=45) | All Subjects (N=225)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 2 | 6
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Haemorrhagic ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Hepatitis B reactivation (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 4
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Meningitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Perihepatic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 4 | 6 | 0 | 4 | 1 | 3 | 2 | 21
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 4
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3
Hepatitis B DNA assay positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 4
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 4
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 5
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EGF816 75 mg (Phase l Part) (N=17) | EGF816 100 mg (Phase l Part) (N=38) | EGF816 150 mg (Phase l Part) (N=73) | EGF816 200 mg (Phase l Part) (N=8) | EGF8166 225 mg (Phase l Part) (N=28) | EGF816 300 mg (Phase l Part) (N=5) | EGF816 350 mg (Phase l Part) (N=11) | EGF816 150 mg (Phase II Part) (N=45) | All Subjects (N=225)
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 10 | 0 | 7 | 3 | 4 | 5 | 35
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 1 | 1 | 0 | 0 | 3 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 7
Angina pectoris (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 3
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 4 | 0 | 1 | 1 | 0 | 2 | 9
Eye discharge (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 5 | 2 | 2 | 0 | 0 | 0 | 9
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 1 | 8
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 4 | 0 | 2 | 0 | 1 | 4 | 16
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 1 | 1 | 2 | 5 | 13
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 4
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 10 | 17 | 1 | 4 | 0 | 0 | 8 | 42
Diarrhoea (Gastrointestinal disorders) | 4 | 13 | 29 | 4 | 17 | 5 | 9 | 21 | 102
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 5 | 0 | 2 | 1 | 0 | 0 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 5 | 0 | 3 | 1 | 1 | 4 | 15
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 5
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 4 | 0 | 1 | 1 | 0 | 2 | 11
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 4
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 8 | 15 | 2 | 10 | 2 | 3 | 10 | 54
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Stomatitis (Gastrointestinal disorders) | 8 | 9 | 20 | 3 | 11 | 1 | 3 | 12 | 67
Vomiting (Gastrointestinal disorders) | 6 | 6 | 10 | 0 | 8 | 1 | 2 | 5 | 38
Asthenia (General disorders) | 1 | 1 | 5 | 0 | 1 | 1 | 1 | 3 | 13
Chest discomfort (General disorders) | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 3 | 9
Chills (General disorders) | 0 | 4 | 2 | 0 | 1 | 0 | 2 | 0 | 9
Early satiety (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 8 | 8 | 21 | 3 | 8 | 3 | 3 | 5 | 59
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3
Influenza like illness (General disorders) | 0 | 2 | 3 | 1 | 2 | 0 | 0 | 1 | 9
Non-cardiac chest pain (General disorders) | 1 | 2 | 10 | 0 | 2 | 0 | 0 | 3 | 18
Oedema peripheral (General disorders) | 1 | 5 | 11 | 2 | 1 | 2 | 0 | 5 | 27
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Pyrexia (General disorders) | 0 | 3 | 8 | 1 | 6 | 2 | 2 | 12 | 34
Swelling face (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Xerosis (General disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 5
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 4
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Conjunctivitis (Infections and infestations) | 0 | 3 | 2 | 1 | 1 | 0 | 0 | 3 | 10
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 4 | 10
Herpes zoster reactivation (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Nasopharyngitis (Infections and infestations) | 2 | 4 | 5 | 1 | 4 | 0 | 0 | 6 | 22
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Paronychia (Infections and infestations) | 1 | 3 | 12 | 2 | 4 | 1 | 4 | 5 | 32
Pharyngitis (Infections and infestations) | 1 | 2 | 2 | 1 | 1 | 0 | 0 | 1 | 8
Pneumonia (Infections and infestations) | 0 | 2 | 4 | 0 | 2 | 1 | 1 | 2 | 12
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 2 | 7
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3
Skin infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 4
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 9 | 7 | 3 | 7 | 0 | 2 | 7 | 36
Urinary tract infection (Infections and infestations) | 2 | 3 | 4 | 2 | 1 | 0 | 0 | 7 | 19
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 4
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 5
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 0 | 3 | 0 | 1 | 2 | 10
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
Alanine aminotransferase increased (Investigations) | 2 | 4 | 4 | 0 | 2 | 0 | 1 | 4 | 17
Amylase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 6 | 9
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 5 | 0 | 3 | 0 | 1 | 5 | 18
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 6
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 5
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 1 | 0 | 4 | 0 | 0 | 1 | 8
Blood creatinine increased (Investigations) | 1 | 2 | 5 | 1 | 4 | 1 | 1 | 1 | 16
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 5
Gamma-glutamyltransferase increased (Investigations) | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 3 | 8
Lipase increased (Investigations) | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 6 | 11
Neutrophil count decreased (Investigations) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 6
Platelet count decreased (Investigations) | 1 | 0 | 3 | 0 | 4 | 1 | 0 | 3 | 12
Weight decreased (Investigations) | 1 | 2 | 3 | 0 | 4 | 0 | 2 | 1 | 13
Decreased appetite (Metabolism and nutrition disorders) | 5 | 4 | 16 | 2 | 7 | 2 | 5 | 13 | 54
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3 | 4 | 0 | 1 | 0 | 1 | 1 | 11
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 3 | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 5 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 9 | 0 | 3 | 0 | 0 | 7 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 11 | 2 | 5 | 1 | 1 | 4 | 34
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 6 | 11 | 3 | 1 | 1 | 0 | 3 | 26
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1 | 2 | 0 | 1 | 1 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 7 | 5 | 0 | 0 | 0 | 0 | 4 | 17
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 6 | 1 | 3 | 0 | 2 | 1 | 16
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 2 | 8
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 6 | 8 | 0 | 2 | 0 | 0 | 3 | 20
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 5
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Aphasia (Nervous system disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 4
Ataxia (Nervous system disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 4
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Dementia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 6 | 9 | 1 | 4 | 2 | 1 | 4 | 32
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 4 | 7
Headache (Nervous system disorders) | 1 | 7 | 13 | 3 | 6 | 1 | 1 | 9 | 41
Hyperaesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 4
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 6
Paraesthesia (Nervous system disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 5
Petit mal epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 5
Taste disorder (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 4
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 6
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 5
Insomnia (Psychiatric disorders) | 2 | 2 | 8 | 3 | 2 | 0 | 0 | 5 | 22
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 4
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 4
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 4
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 21 | 3 | 10 | 2 | 2 | 14 | 64
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 13 | 0 | 8 | 1 | 1 | 6 | 36
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 2 | 0 | 1 | 2 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 6 | 0 | 2 | 2 | 0 | 0 | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 5 | 1 | 2 | 1 | 3 | 1 | 16
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 6
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 3 | 0 | 0 | 3 | 9
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 2 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 2 | 8
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 8 | 2 | 6 | 0 | 0 | 1 | 19
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 5 | 9
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 4 | 8 | 1 | 5 | 0 | 3 | 10 | 34
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 9 | 15 | 1 | 11 | 3 | 5 | 5 | 52
Eczema (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 2 | 1 | 0 | 0 | 1 | 10
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 11 | 28 | 5 | 12 | 3 | 6 | 13 | 82
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 4 | 0 | 2 | 1 | 2 | 8 | 24
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 5
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 5 | 0 | 4 | 2 | 0 | 2 | 15
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 9 | 29 | 4 | 15 | 5 | 6 | 17 | 89
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 3 | 0 | 0 | 1 | 8
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 5
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 3 | 1 | 0 | 1 | 8
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1 | 5 | 1 | 4 | 0 | 2 | 3 | 19
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 4 | 2 | 1 | 2 | 0 | 1 | 8 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT02108964/Prot_002.pdf
  • Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT02108964/SAP_003.pdf